CLINICAL TRIAL: NCT06473194
Title: Physiological and Biochemical Effects of Laparoscopic Anesthesia and Surgery
Brief Title: This Study Assess Some Physiological Parameters, Blood Picture, and Hemodynamic Parameters, Blood Pressure, Respiratory Assess by SPO2, During Different Periods in Laparoscopic Surgery
Acronym: laparoscopy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mohammed Abdulhameed (Other)
Responsible Party: Sponsor-Investigator, Mohammed Abdulhameed, principal investigator, Tunis University
Organization: Tunis University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: physiological measurement
Record Dates: First submitted 2024-06-01; First posted 2024-06-25 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-06

CONDITIONS: Anesthesia Complication; Physiological Parameter
MeSH Terms: interventions — Rocuronium; Heart Rate; Oxygen Saturation

STUDY DESIGN:
Intervention Model Description: describe techniques of laparoscopic procedures. 2. Discuss complications and assessments of patients who undergo laparoscopic procedures. 3. to assess liver function and hematological effects due to laparoscopic surgery 4. cardiovascular and respiratory squeal due to laparoscopic complication is minor compared to open surgery and can be managed rapidly.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- age , gender (Experimental): group according to age and according to gender
  Interventions: Procedure: general anesthesia drug (like Propofol, esmeron, and ketamin, .effects of pneumoperitoneum

INTERVENTIONS:
Procedure: general anesthesia drug (like Propofol, esmeron, and ketamin, .effects of pneumoperitoneum — this research will involve the selection of elective cases with ASA class I or II and assessment of patients with respiratory cardiovascular parameters and hematology perioperative
  Other Names: monitoring in anesthesia to asses hemodynamic parameter includes blood pressure, pulse rate, and SPO2, compared with biochemical blood sugar, liver enzyme, respiratory alteration by end-tidal CO2

SUMMARY:
Laparoscopic surgery is widely used now. These benefits included many items, e.g. reducing post-operative pain, cosmetic the result was improved, and the patient also had more satisfaction for the patient and reduced hospital stay. This surgery involved insufflation of gas into the peritoneal cavity, producing pneumoperitoneum, and causing an increase in intra-abdominal pressure. The raised intraabdominal pressure of the pneumoperitoneum, the patient's position alteration, and the absorption of carbon dioxide into the abdomen have a direct effect on causing a change in physiology, especially in the cardiovascular and respiratory systems. These effects, as well as a direct effect of gas insufflation, may have significant effects on the patient especially if the patient has a comorbidity or is elderly.

DETAILED DESCRIPTION:
The objective of this study was to assess the technique used in laparoscopic surgery and their associated complications, including some hematological parameters, (these include blood pictures and liver enzymes), respiratory, (including the inspired and expired tidal volume, oxygen saturation, airway pressure, plateau pressure, and use of PEEP) cardiovascular system (including the systolic, diastolic, and mean blood pressure, heart rate)

ELIGIBILITY:
Inclusion Criteria:

1. elective abdominal surgery
2. a healthy, fit person
3. use of general anesthetics
4. use of pneumoperitoneum and CO2 insufflation

Exclusion Criteria:

1. emergency condition
2. patient with cardiovascular disease

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
blood pressure. | during preoperative, 5 minute, intraoperative every five minute with post operative read after one hour
  blood pressure in mmHg, pulse rate in beat per minute
AST and ALT liver enzymes were measured, by blood samples taken intravenously in the perioperative period | 5 minute pre-operation and 5 minute postoperative
  in unit/liter
blood sugar, should measured and assessed with different groups | 5 minute during pre-operative and 15 minute post- operative period
  blood sugar in mg/dl
end-tidal Co2, measured and compared statistically with other parameter | perioperatively every 5 minute
  End-tidal Co2 in CMH2O
pulse rate measured continuously during intra-operative and compared with other hemodynamic parameter | 5 minute during preoperative, and continue every 5 minute in perioperatively
  beat per minute (BPM)

SECONDARY OUTCOMES:
measurement of body weight | measured preoperative period by 5 minute and post-operative during 15 minute
  in Kg

CONTACTS AND LOCATIONS:
Overall Officials: hussam Mu. Kareem, PHD, Study Director — Ministry of Health

IPD SHARING:
Plan to Share IPD: No
after approval and acceptance these data would be available soon

REFERENCES:
- [Background] Celep RB, Kahramanca S, Ozsoy M, Azili C, Cetinkunar S, Hasdemir AO, Guzel H, Ozgehan G, Colhan I, Kucukpinar TH. Effects of intraabdominal pressure on mean platelet volume during laparoscopic cholecystectomy. Turk J Med Sci. 2014;44(3):360-4. doi: 10.3906/sag-1304-23. PMID 25558633
- [Background] Bitkin A, Aydin M, Irkilata L, Keles M, Akgunes E, Ocak S, Atilla MK. Effect of Intra-abdominal Pressure Rise on Hematological Parameters in Laparoscopic Urologic Surgery. J Coll Physicians Surg Pak. 2018 Sep;28(9):699-702. doi: 10.29271/jcpsp.2018.09.699. PMID 30158037
- [Background] Sen MC, Turkyilmaz Z, Sonmez K, Karabulut R, Kaya Z, Yenicesu I, Gursel T, Basaklar AC. The Effect of Carbon Dioxide Insufflation Applied at Different Pressures and Periods on Thrombotic Factors. Indian J Hematol Blood Transfus. 2016 Mar;32(1):87-91. doi: 10.1007/s12288-015-0517-2. Epub 2015 Feb 15. PMID 26855512
- [Background] Crema E, Ribeiro EN, Hial AM, Alves Junior JT, Pastore R, Silva AA. Evaluation of the response of cortisol, corticotropin and blood platelets kinetics after laparoscopic and open cholecystectomy. Acta Cir Bras. 2005 Sep-Oct;20(5):364-7. doi: 10.1590/s0102-86502005000500005. Epub 2005 Sep 5. PMID 16186960
- [Background] Hasukic S, Kosuta D, Muminhodzic K. Comparison of postoperative hepatic function between laparoscopic and open cholecystectomy. Med Princ Pract. 2005 May-Jun;14(3):147-50. doi: 10.1159/000084630. PMID 15863986